CLINICAL TRIAL: NCT02312843
Title: A Randomized Controlled Trial to Examine the Effects of Aerobic Exercise on Cognition and Aging-related Biomarkers for Adults With Prediabetes and Mild Cognitive Impairment
Brief Title: Piedmont Aging, Cognition & Exercise Study-2
Acronym: PACE-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00022598
Record Dates: First submitted 2014-10-03; First posted 2014-12-09 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Mild Cognitive Impairment; Prediabetes
Keywords: Mild Cognitive Impairment; Cognitive disorders; Prediabetes; Exercise
MeSH Terms: conditions — Cognitive Dysfunction; Prediabetic State; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Intensity Program-aerobic exercises (Active Comparator): This exercise program will consist of walking or running on a treadmill or elliptical trainer, or spinning on a stationary bicycle. The goal of the program will be for participants to exercise at a moderate to high level of intensity, defined as 70-80% (American College of Sports Medicine guidelines) of heart rate reserve (HRR), for 45-60 minutes 4 days per week. At the start of each training session and following a 5-minute warm-up, subjects will exercise at 50% HRR (0.5[HRmax-HRrest] +HRrest) and intensity will gradually be increased to the individualized target heart rate training zone. Exercise facilitators will use a pre-specified computerized program. This program provides guidelines for the individualized progression of exercise based on age and resting heart rate. Subjects will wear a digital heart rate monitoring device for the duration of the training session to ensure they are exercising safely at the specified level of intensity.
  Interventions: Behavioral: Exercise/Aerobic
- Low-intensity Program-Stretching (Placebo Comparator): The low-intensity activity program will consist of an individualized and organized series of stretching and balance activities for the whole body, specifically designed for older adults. Consistent with the high-intensity protocol, subjects will complete the prescribed 45-60 minute stretching routine 4 days per week at the exercise facility. All stretching routines will include warm-up and cool-down activities, and will be within each subject's range of motion. Each stretch will be held for 20-30 s and repeated 5-10 times. Subjects will wear a digital heart rate monitoring device to ensure they are stretching safely and at an intensity below 35% HRR. The activity log completed during each stretching session will include HR, stretching duration, and mean HR during stretching. Subjects will also have the option to participate in structured pre-approved (by the exercise facilitator) stretching classes at the exercise facility when available.
  Interventions: Behavioral: Exercise/Stretching

INTERVENTIONS:
Behavioral: Exercise/Aerobic
  Arms: High-Intensity Program-aerobic exercises
Behavioral: Exercise/Stretching
  Arms: Low-intensity Program-Stretching

SUMMARY:
The purpose of this research study is to examine the effects of high and low intensity exercise for those with mild memory loss and pre-diabetes. The investigators will also examine the effects of this exercise on certain proteins and hormones in body fluids, and on brain structure and function using magnetic resonance imaging (MRI). Recent studies indicate that exercise improves memory and thinking abilities for adults with mild memory loss OR pre-diabetes. This study examines the effects of exercise on people with mild memory loss AND pre-diabetes.

ELIGIBILITY:
Inclusion Criteria:

* 50 years or older
* Mild memory concerns
* In good health
* Not taking diabetes medications
* Not currently exercising

Exclusion Criteria:

* Significant neurologic disease that might affect cognition, such as AD, stroke, Parkinson's disease, multiple sclerosis, or severe head injury with loss of consciousness > 30 min or with permanent neurologic sequelae;
* Significant medical illness or organ failure, such as:
* Liver disease: history of hepatitis or hepatic failure
* Significant elevations in liver function tests: lab values more than 2.5 times the upper limit of normal
* Kidney disease known history of kidney failure.
* Uncontrolled hypertension
* Cardiovascular disease, defined as: any acute cardiovascular abnormality, such as new or unstable angina, uncontrolled irregular heart beat (treated a-fib and occasional PVC's are OK) or symptomatic heart failure, acute shortness of breath for any reason, or clinically significant edema, is an exclusion. History in the last year of myocardial infarction, angina, coronary artery angioplasty, bypass grafting, pacemaker insertion, STENT placement, postural hypotension, transient ischemic attack, or carotid artery surgery.
* Chronic lung disease, such as: COPD/emphysema
* Hemoglobin A1c levels that fall outside the range of 5.7-6.4%; If 2-h OGTT glucose values 220 mg/dL and hemoglobin A1c levels meet inclusion criteria (5.7-6.4%), then PCP written indication that no pharmacologic intervention for type 2 diabetes is needed at present will be required for continued study participation.
* Current use of anti-psychotic, anti-convulsant, anxiolytic, or sedative medication;
* Current use of any cognition-enhancing medication, including experimental medications within the past 60 days;
* Current or previous use of hypoglycemic agents or insulin (except during pregnacy); diabetics previously on oral agents but have been off of them for > 1 year are ok pending PI and study physician approval.
* Musculoskeletal impairment sufficient to interfere with study participation

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-03; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in cognitive performance from baseline following 6 month of high or low intensity exercise regimen | 2 assessments, one before and one after 6 months of exercise
  The cognitive variables identified above, by domain, will be subjected to separate treatment group X treatment month (3, 6) multivariate analyses of covariance (MANCOVA), with baseline scores and age serving as covariates. When the MANCOVA proves significant, separate post-hoc analysis of covariance (ANCOVA) will be conducted on the relevant dependent variables.
  Cognitive tests include measures of executive function and working memory.

SECONDARY OUTCOMES:
Change from baseline in blood sugar concentration and cerebrospinal fluid glucose measures during an oral glucose tolerance test following 6 months of high or low intensity exercise | 3 Oral glucose tolerance tests over a 6 month period; 2 lumbar punctures, one before and one after the 6 month exercise regimen
  Multiple regression and correlational (MRC) analyses will be conducted to evaluate whether treatment-induced change in insulin sensitivity and in other blood and cerebrospinal fluid biomarkers predict cognitive performance among subjects in the aerobic group.

OTHER OUTCOMES:
Change from baseline in brain network connectivity using brain imaging | 2 brain scans over a 6 month period, one before and one after the 6 month exercise regimen
  Whole-brain averages will be computed, reflecting characteristics of the entire system. Whole-brain averages will be compared with random networks generated with the same node number and degree,48 and will be compared between intervention groups using general linear regression models. Regions of interest (hippocampus, posterior cingulate/precuneus, prefrontal cortex) will be extracted using WFU Pickatlas and regional degree, Eglob, or Eloc will be compared between groups using the general linear model.

CONTACTS AND LOCATIONS:
Overall Officials: Laura D. Baker, Ph.D, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States